CLINICAL TRIAL: NCT07307118
Title: Functional Hip Strength and Pain Changes in Women With Knee Osteoarthritis Following a Single-Dose Intra-Articular Platelet-Rich Plasma Injection and a 6-Week Home Exercise Program: A Single-Group Longitudinal Study
Brief Title: Functional Hip Strength Improvement in Knee Osteoarthritis Following Single-Dose PRP and a 6-Week Home Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Muharrem Gökhan Beydağı, Assistant Professor, Firat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FU_MGBeydagi_PRP_B_2025/12/150
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis (OA)
Keywords: Knee osteoarthritis; exercise therapy; hip muscle strength; platelet-rich plasma; Hand-held dynamometer; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group: PRP Injection + Home Exercise Program (Experimental): All participants received a unilateral single-dose intra-articular platelet-rich plasma (PRP) injection for symptomatic knee osteoarthritis, followed by a 6-week home-based strengthening and functional exercise program performed 3 times per week. The exercise program targeted knee extensors/flexors and hip extensors/abductors/external rotators. Participants were encouraged to walk at least 30 minutes on at least 5 days per week and were contacted weekly by phone to support adherence.
  Interventions: Biological: Platelet-Rich Plasma (PRP) Injection; Behavioral: Home Exercise Program

INTERVENTIONS:
Biological: Platelet-Rich Plasma (PRP) Injection — A single unilateral intra-articular autologous platelet-rich plasma (PRP) injection was administered to the affected knee. Baseline assessments were conducted 5 days following the injection.
  Other Names: PRP
Behavioral: Home Exercise Program — Home-based exercise program performed 3 times per week for 6 weeks, designed to strengthen knee extensors/flexors and hip extensors/abductors/external rotators. Exercises included: quadriceps strengthening (supine isometric contractions with 5-second hold; seated knee extension with 5-second hold; straight leg raise with 5-second hold), hamstring strengthening (supine isometric contractions with 5-second hold; prone active knee flexion with 5-second hold), hip stabilizer strengthening (clamshells and side-lying hip abduction with 5-second hold), and functional exercises (step-ups, forward touchdowns from a step, side stepping, sit-to-stand from a chair without using arms, and partial wall squats), typically 10-15 repetitions. Participants were also encouraged to walk at least 30 minutes on at least 5 days per week, and adherence was supported via weekly telephone contact.

SUMMARY:
This single-group longitudinal study evaluated changes in hip stability isometric strength, knee muscle strength, and activity-related pain in women with knee osteoarthritis following a single-dose intra-articular platelet-rich plasma (PRP) injection and a 6-week home exercise program. Outcomes were assessed at baseline (5 days post-injection), week 6, and week 12. The intervention included strengthening exercises for knee and hip muscle groups performed three times per week and regular walking encouragement with weekly phone follow-up for adherence.

DETAILED DESCRIPTION:
Participants with unilateral symptomatic knee osteoarthritis performed a standardized 6-week home strengthening program (knee extensors/flexors; hip extensors/abductors/external rotators) three times weekly and were encouraged to walk regularly. Hip Stability Isometric Test (HipSIT), quadriceps/hamstring strength (hand-held dynamometry, normalized to body mass), and activity pain (VAS 0-10) were measured at baseline, week 6, and week 12 to evaluate functional strength and symptom changes after PRP plus exercise.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 45-70 years.
* Radiographic knee osteoarthritis: Kellgren-Lawrence grade II-III in the affected knee and grade II or less in the unaffected knee.
* Unilateral knee pain during activity with VAS score ≥5 (for at least the past 3 months).
* Referred to physiotherapy following a unilateral single-dose PRP injection.

Exclusion Criteria:

* Any intra-articular knee injection within the past 6 months.
* Regular lower-extremity strengthening exercise or non-pharmacological treatment for knee OA within the past 6 weeks.
* History of lower-extremity surgery.
* History of neurological, rheumatological and/or cognitive diseases.
* Unable to use a telephone.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2025-07-08 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-13 (Actual)

PRIMARY OUTCOMES:
Hip Stability Isometric Test (HipSIT) strength (N/kg), affected side | Baseline (5 days post PRP injection), Week 6, Week 12
  Hip stability isometric strength (combined hip extensor, abductor and external rotator maximum isometric strength) assessed using a hand-held dynamometer during the Hip Stability Isometric Test (HipSIT). The test is performed in side-lying "clam" position (hip 45° flexion, knee 90° flexion). Three maximal trials (5 seconds each) are performed and the maximum force output (N) is normalized to body mass (N/kg).

SECONDARY OUTCOMES:
Quadriceps femoris isometric strength (N/kg), affected side | Baseline (5 days post PRP injection), Week 6, Week 12
  Maximum isometric quadriceps strength measured with a hand-held dynamometer in sitting position (hip 90° flexion, knee semi-flexion), with the dynamometer placed on the anterior surface of the ankle. Three maximal trials (5 seconds each) are performed and the maximum force output (N) is normalized to body mass (N/kg).
Hamstring isometric strength (N/kg), affected side | Baseline (5 days post PRP injection), Week 6, Week 12
  Maximum isometric hamstring strength measured with a hand-held dynamometer in prone position (hip neutral, knee flexion 90°), with the dynamometer placed on the proximal posterior surface of the ankle. Three maximal trials (5 seconds each) are performed and the maximum force output (N) is normalized to body mass (N/kg).
Knee pain during activity (Visual Analog Scale, 0-10) | Baseline (5 days post PRP injection), Week 6, Week 12
  Pain severity during activity assessed using a 10-cm Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain).

OTHER OUTCOMES:
Strength symmetry indices (QI, HI, HipI), % | Baseline (5 days post PRP injection), Week 6, Week 12
  Strength symmetry indices calculated as (affected side isometric strength / unaffected side isometric strength) × 100 for HipSIT (HipI), quadriceps (QI), and hamstrings (HI).

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat Üniversitesi, Elâzığ, MErkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No